CLINICAL TRIAL: NCT03684356
Title: Comparison of the Dimensional Changes of Hard and Soft Peri-implant Tissues Around Single Immediate Post-Extraction Implants in the Esthetic Zone With Socket Shield Technique Versus Using Xenograft: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Peri-implant Tissues Using Socket Shield Technique Versus Xenograft
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Atef Abd El Moneium, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU12
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Socket Shield
MeSH Terms: interventions — Immediate Dental Implant Loading; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): immediate implant with socket shield technique
  Interventions: Procedure: socket shield technique
- control (Active Comparator): immediate implant placement with filling the buccal gap with xenograft
  Interventions: Procedure: xenograft

INTERVENTIONS:
Procedure: socket shield technique — immediate implant placement with buccal part of the root is retained
  Arms: experimental
Procedure: xenograft — immediate implant placement with filling the buccal gap with xenograft
  Arms: control

SUMMARY:
The aim of this study is to clinically and radiographically evaluate the dimensional changes of soft and hard peri-implant tissues around single immediate post-extraction implants in the esthetic zone.

DETAILED DESCRIPTION:
to compare the efficacy of the socket shield technique in counteracting the dimensional changes of the soft and hard peri-implant tissues to filliing the buccal gap with xenograft.

* Population (P): Patients with single non-restorable tooth in the esthetic zone.
* Intervention (I): Immediate implant placement with socket shield technique.
* Comparator (C): Immediate implant placement and filling the buccal gap with xenograft.
* Primary Outcome (O): Pink Esthetic Score (PES) (Fürhauser et al., 2005).
* Time frame: 9 months (Chu et al., 2015).
* Study design: Randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age was 18 years or older.
2. Non-restorable tooth in the upper inter-bicuspid area.
3. Adequate bone volume for the placement of immediate implant.
4. Following tooth extraction, there was an intact socket bony wall (type I extraction socket).
5. Primary stability of the implant was achieved at the time of the implant placement.

Exclusion Criteria:

1. Patients who reported tobacco use in the past 5 years.
2. Patients who had severe periodontal destruction at the site of implant placement.
3. The presence of any signs of acute infection in the surgical site or the adjacent two natural teeth.
4. Patients who had history of any systemic disease that precludes the placement of implants.
5. Any disease that might affect bone metabolism as osteoporosis.
6. Patients taking medications that might affect bone turn over as bisphosphonates.
7. Physically or mentally handicapped patients.
8. Pregnant females.
9. Teeth with vertical root fractures on the buccal aspect
10. Teeth with any other pathologies affecting the buccal part of the root, for example, external or internal resorptions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
pink esthetic score | 9 months
  Pink esthetic score evaluates the soft tissue esthetics around implant supported crowns. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value. The maximum achievable PES is 14. 7 variables are measured: mesial and distal papillae being 0 if absent, 1 if incomplete and 2 if complete. Alveolar process, soft tissue level, contour, texture and color being 0 if major discrepancy, 1 if minor discrepancy and 2 if matches the contralateral

SECONDARY OUTCOMES:
Recession of the buccal peri-implant mucosa | 9 months
  measured at the apical zenith of the mucosal margin on the implants after digital superimposition of the optically scanned models as the vertical distance change between the former and the new position of soft tissue margins.
Corono-apical peri-implant bone dimensional changes | 6 months
  measured at the middle of the buccal implant surface after the superimposition of Cone Beam C.T scans as the difference between the former and new vertical distance from the implant platform to the buccal alveolar crest
Bucco-lingual peri-implant bone dimensional changes | 6 months
  measured at middle of the buccal implant surface 1mm below the alveolar crest after the superimposition of the Cone Beam C.T scans as the difference between the former and new horizontal distance between the buccal and the palatal plate of bone
Patient satisfaction: VAS | 9 months
  Patient satisfaction will be evaluated using a questionnaire which is based on a visual analog scale (VAS). A horizontal VAS bar, 100 mm long, with the right anchor labeled "much less than natural teeth" which is marked by zero and the left anchor labeled "much more" which is marked by 10 will be used. Five questions will be formulated to record the patients' satisfaction in terms of functionality and from an esthetic point of view. Participants will look in a mirror and also be viewed a photograph before recording their answers on the horizontal calibrated line.

CONTACTS AND LOCATIONS:
Overall Officials: Amr F Zahran, Professor, Study Chair — Professor in Department of Oral Medicine and Periodontology
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumer D, Zuhr O, Rebele S, Hurzeler M. Socket Shield Technique for immediate implant placement - clinical, radiographic and volumetric data after 5 years. Clin Oral Implants Res. 2017 Nov;28(11):1450-1458. doi: 10.1111/clr.13012. Epub 2017 Mar 23. PMID 28333394
- [Background] Bramanti E, Norcia A, Cicciu M, Matacena G, Cervino G, Troiano G, Zhurakivska K, Laino L. Postextraction Dental Implant in the Aesthetic Zone, Socket Shield Technique Versus Conventional Protocol. J Craniofac Surg. 2018 Jun;29(4):1037-1041. doi: 10.1097/SCS.0000000000004419. PMID 29489581
- [Background] Mitsias ME, Siormpas KD, Kotsakis GA, Ganz SD, Mangano C, Iezzi G. The Root Membrane Technique: Human Histologic Evidence after Five Years of Function. Biomed Res Int. 2017;2017:7269467. doi: 10.1155/2017/7269467. Epub 2017 Nov 22. PMID 29333449
- [Background] Siormpas KD, Mitsias ME, Kontsiotou-Siormpa E, Garber D, Kotsakis GA. Immediate implant placement in the esthetic zone utilizing the "root-membrane" technique: clinical results up to 5 years postloading. Int J Oral Maxillofac Implants. 2014 Nov-Dec;29(6):1397-405. doi: 10.11607/jomi.3707. Epub 2014 Sep 26. PMID 25265125
- [Background] Tan Z, Kang J, Liu W, Wang H. The effect of the heights and thicknesses of the remaining root segments on buccal bone resorption in the socket-shield technique: An experimental study in dogs. Clin Implant Dent Relat Res. 2018 Jun;20(3):352-359. doi: 10.1111/cid.12588. Epub 2018 Feb 8. PMID 29417708
- [Derived] Atef M, El Barbary A, Dahrous MSE, Zahran AF. Comparison of the soft and hard peri-implant tissue dimensional changes around single immediate implants in the esthetic zone with socket shield technique versus using xenograft: A randomized controlled clinical trial. Clin Implant Dent Relat Res. 2021 Jun;23(3):456-465. doi: 10.1111/cid.13008. Epub 2021 May 24. PMID 34028974